CLINICAL TRIAL: NCT05473403
Title: Validation of a Prognostic Score for Steroid Therapy Response in Acute Severe Autoimmune Hepatitis, a National Prospective Multicentre Study
Brief Title: Validation of a Prognostic Score for Steroid Therapy Response in Acute Severe Autoimmune Hepatitis
Acronym: PRO-SURFASA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D20180121; 2021-A01869-32 (Other: IDRCB)
Record Dates: First submitted 2022-06-07; First posted 2022-07-25 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-09

CONDITIONS: Liver Failure, Acute; Hepatitis, Autoimmune; Organ Dysfunction Scores; Risk Factors
Keywords: Acute Severe AutoImmune Hepatitis (ASAIH); Decisional score; Prognostic score
MeSH Terms: conditions — Liver Failure, Acute; Hepatitis, Autoimmune

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prognostic, non-randomized, comparative, longitudinal, prospective, external validation cohort, which aims to evaluate a decisional score previously developed in a retrospective cohort.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid therapy (Experimental): Prednisone or Prednisolone or Methylprednisolone : Patient with ASAIH will be treated in oral or intravenous (IV) with high doses ( ≥ 1mg/kg/day) of corticosteroids (Prednisone or Prednisolone or Methylprednisolone) until relapse (confirmed by blood tests and clinical status) requiring an emergency Liver Transplantation (LT) or death.
  Interventions: Other: Corticosteroid therapy
- Patient without corticosteroid therapy (No Intervention): Patient not treated will undergo to emergency Liver Transplantation (LT) or death.

INTERVENTIONS:
Other: Corticosteroid therapy — Administration of high doses of corticosteroids as early as possible. Patient non-responder to treatment should lead to listing for emergency liver transplantation (LT).
  Arms: Corticosteroid therapy

SUMMARY:
Autoimmune hepatitis (AIH) is a chronic liver disease, which is characterized by the increase of immunoglobulin G (IgG) level, the presence of auto-antibodies and a typical histology, in the absence of other liver disease.

Due to the heterogeneity of AIH manifestations, different scoring systems have been validated in order to make a reliable diagnosis. The two most recent scoring systems are: the revised International Autoimmune Hepatitis Group (IAIHG) criteria and the IAIHG simplified criteria. The second one is recommended by the European Association for the Study of the Liver (EASL) clinical practice guidelines (CPGs).

The EASL clinical practice guidelines suggests that the treatment of ASAIH (Acute Severe AIH) is high doses of corticosteroids (superior to 1mg/kg/day) as early as possible and a lack of improvement within seven days should lead to listing for emergency liver transplantation (LT). However, the "lack of improvement" is not objectively defined and the grading of recommendation is III (Opinions of respected authorities).

The hypothesis of the study is that the previously developed decisional score on a retrospective series will prospectively allow the differentiation between patients with ASAIH (Acute Severe AIH) who respond to corticosteroid therapy and should be maintained on treatment and patients who do not respond and should be rapidly evaluated for LT. The score will be computed at day 3 since corticosteroid introduction.

DETAILED DESCRIPTION:
All the interventions (blood samples, imagery examinations, visits, liver biopsy, corticosteroid therapy, liver transplantation) will be performed following the standard of care for ASAIH. The investigators of the participating centers will not change their standard management for the study protocol. The management will follow the recommendation of EASL CPGs.

The prognostic score will allow to distinguish between patient's responders and non-responders to corticosteroid therapy in ASAIH. This knowledge will avoid the prolonged duration of the corticosteroid therapy in patients for whom this therapy is futile or harmful and rapidly select the patients for LT. Of course considering that the created score is decisional whether a patient is a candidate for LT, a prospective validation is mandatory to use it as a clinical tool for the day-to-day practice. This is the first prospective study on ASAIH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Strong clinical suspicion of severe acute autoimmune hepatitis defined by the presence of increased IgG and/or autoantibodies and/or histology characteristic of the disease in the absence of other causes of severe acute hepatitis.
* International Normalized Ratio (INR) ≥ 1.5
* Informed, written consent
* Patient having the rights to French social insurance

Exclusion Criteria:

* Previous medical history of chronic liver disease including autoimmune liver disease (AIH, Primary Biliary Cholangitis (PBC), Primary Sclerosing Cholangitis (PSC) , alcoholic hepatitis etc.)
* Other causes of acute severe hepatitis:

  * Hepatitis A Virus (HAV) hepatitis, defined by HAV Immunoglobulin M (IgM) antibodies
  * Hepatitis B Virus (HBV) hepatitis, defined by HBs antigen and HBV IgM antibodies
  * Hepatitis E Virus (HEV) hepatitis, defined by HEV IgM antibodies or positive HEV-RNA in immunosuppressed patients
  * Drug induced hepatitis, histologically proved or induced by well-known hepatotoxic substances
  * Acute hypoxemic hepatitis, context of shock, hypoxemia or heat shock
  * Budd-Chiari syndrome, diagnosed by imagery (Doppler ultrasound, CT scan)
  * Acute hepatitis in the context of a HELLP (Hemolysis, Elevated Liver enzymes and a Low Platelet count) syndrome or acute fatty liver of pregnancy
* Use of corticosteroids 1 month before inclusion
* Pregnant or lactating woman
* Curator or guardianship or patient placed under judicial protection
* Participation in other interventional research during the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Prospectively validate the previously elaborated SURFASA-score, evaluating its ability to predict non-response outcome to corticosteroid therapy in a new population of patients with acute severe autoimmune hepatitis. | Day 90
  Patient response within 90 days to corticosteroid therapy defined as: responders (alive without LT) or non-responders (dead or transplanted) within 90 days since corticosteroid therapy introduction.

SECONDARY OUTCOMES:
The association between infection occurrence and death during hospitalization | participation period (treatment+follow-up): 12 months
  Documented infections during hospitalization
the management of infected ASAIH patients in usual practice | participation period (treatment+follow-up): 12 months
  Antibiotic therapy : doses
The risk factors for early AIH flair after corticosteroid therapy response. | D90
  The frequency of AIH flair
The risk factors for AIH recurrence after liver transplantation | participation period (treatment+follow-up): 12 months
  AIH recurrence
The evolution of patients after LT | participation period (treatment+follow-up): 12 months
  Retransplantation, alive, death
The evolution of patients not treated with corticosteroids but meeting the inclusion and non-inclusion criteria | participation period (treatment+follow-up): 12 months
  Retransplantation, alive, death
The prognostic factors for survival in patients treated with corticosteroids who underwent or not LT | participation period (treatment+follow-up): 12 months
  quality of the graft, immunosuppression, rejection episode,
The association of histological features (liver biopsy) with response to corticosteroids and survival at 90 days since admission | 90 days
  Presence of centrilobular necrosis and inflammatory infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora DE MARTIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (26):
- France (26):
  - CHU Angers, Service Hepato-gastro-enterologie, Angers
  - CHU Jean Minjoz Besançon, Service d'hepatologie et de soins intensifs digestifs, Besançon
  - APHP, Hopital Avicenne, Service Hepatologie et Oncologie Hépatique, Bobigny
  - CHU Brest, Hopital de la Cavale Blanche Service Gastro-enterologie, Brest
  - CHU de Caen, Hopital de la Cote de Nacre, Service Hepato-Gastro-Enterologie et Nutrition, Caen
  - CHU Trousseau Chambray, Service Gastro-enterologie et hepatologie, Chambray-lès-Tours
  - CHU Dijon, Service Hepato-gastroenterologie et cancerologie digestive, Dijon
  - CHRU de Lille, Hopital Claude Huriez, Service des maladies de l'appareil digestif et de la nutrition, Lille
  - CHU Limoges, Hopital Dupuytren, Service Hepato-gastroenterologie et nutrition, Limoges
  - CHU Hopital Edouard Herriot, Service Hepato-gastro-enterologie, Lyon
  - CHU Lyon, Hopital Croix Rousse, Service Hepato-gastro-enterologie, Lyon
  - Hopital Saint Joseph, Service Hepato-gastro-enterologie, Marseille
  - CHU Montpellier, Hopital Saint Eloi, Service Hepato-gastro-enterologie, Montpellier
  - CHU Nice, Hopital de l'Archet 2, Service Hepatologie, Nice
  - CHU Orleans, Hopital de la Source, Service Gastro-enterologie et hepatologie, Orléans
  - AP-HP, Hopital St Antoine, Service Hepato-gastro-enterologie, Paris
  - APHP, Hopital Pitie-Salpetriere, Service d'hepatologie et de gastroenterologie, Paris
  - AP-HP, Hopital Cochin Service Hepatologie, Paris
  - CHU Bordeaux, GH Sud Haut-Leveque, Service Hepato-gastro-enterologie, Pessac
  - CHU La Miletrie, Service Hepato-gastro-enterologie, Poitiers
  - CHU Reims, Hopital Robert Debré, Service Hepato-Gastroenterologie et de Cancerologie digestive, Reims
  - CHU de Rennes, Hopital de Pontchaillou, Service Maladie du foie, Rennes
  - CHU Rouen, Service d'hepatogastro-enterologie, Rouen
  - CHU Strasbourg, Hopital de Hautepierre, Service Hepato-gastro-enterologie, Strasbourg
  - CHU Toulouse, Hopital Rangueil, Service Hepatologie, Toulouse
  - AP-HP, Paul Brousse Hospital, Centre Hepato-Biliaire, Villejuif

IPD SHARING:
Plan to Share IPD: No